CLINICAL TRIAL: NCT06341023
Title: Functional Balance Intervention (FBI) for Physical and Cognitive Symptoms of Multiple Sclerosis
Brief Title: Functional Balance Intervention in Multiple Sclerosis
Acronym: FBIinMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Tanvi Bhatt, Full professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-1430
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Functional Balance; Cognition; Dual task; Physical function; Muscular strength; Spasticity; Sensorimotor dysfunction; Fall prevention; Vestibular
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be blinded to group existence and assignment and outcome assessors will be blinded to group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lab-based FBI (Experimental): Participants in the lab-based functional balance intervention (FBI) group will receive 4 months of exercise training in the lab (2 times per week for 16 weeks, total 32 sessions). The exercise training will consist of multiple components including functional agility, functional strength, dual-tasking and vestibular exercises.
  Interventions: Behavioral: Functional Balance Intervention
- Lab-based Stretching (Active Comparator): Participants in the lab-based stretching group will receive 4 months of stretching in the lab (2 times per week for 16 weeks, total 32 sessions).The stretching program will include progressive stretches for upper and lower-limb muscles, core and back muscles followed by a cool-down of 10 mins including relaxation and breathing exercises. Stretching exercises will include single and multi-joint stretches designed to target improvements in performance of daily living activities.
  Interventions: Behavioral: Stretching
- Home-based FBI (Experimental): Participants in the home-based functional balance intervention (FBI) group will be asked to complete 4 months of exercise training at home (2 times per week for 16 weeks, total 32 sessions). The exercise training will consist of multiple components including functional agility, functional strength, dual-tasking and vestibular exercises.
  Interventions: Behavioral: Functional Balance Intervention
- Home-Based Stretching (Active Comparator): Participants in the home-based stretching group will be asked to complete 4 months of stretching at home (2 times per week for 16 weeks, total 32 sessions).The stretching program will include progressive stretches for upper and lower-limb muscles, core and back muscles followed by a cool-down of 10 mins including relaxation and breathing exercises. Stretching exercises will include single and multi-joint stretches designed to target improvements in performance of daily living activities.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Functional Balance Intervention — Participants in the intervention group will undergo a multi-component FBI exercise program, both in a lab setting (Study 1) and at home (Study 2), for 2 days/week over 4 months. This evidence-based protocol, previously piloted with chronic stroke patients, older adults with mild cognitive impairment, and pre-frail older adults, focuses on improving physical (endurance, strength, balance, and gait) and cognitive function (processing speed, attention, and memory). The program consists of functional agility, functional strength, dual-task, and vestibular exercises, with each 1-hour session including 10 minutes dedicated to each component. The exercise order will be randomized for each session, preceded by a warm-up with gentle self-stretching exercises.
  Arms: Home-based FBI; Lab-based FBI
Behavioral: Stretching — Participants in the control group will undergo a 4-month lab-based stretching program, with the same frequency and session length as the intervention group (1 hour/session for 2 days/week). The stretching regimen will include progressive stretches targeting upper and lower-limb muscles, core, and back muscles, followed by a 10-minute cool-down comprising relaxation and breathing exercises. These stretches are designed to improve performance in daily living activities. In Study 2, stretching participants will receive a detailed printed exercise manual for home-based training, ensuring consistency with the lab-based program. No additional equipment, such as computers or tablets, is required for the home stretching program.
  Arms: Home-Based Stretching; Lab-based Stretching

SUMMARY:
This project involves two sub-parts:

Study 1: Effect of lab-based Functional Balance Intervention (FBI) for physical and cognitive symptoms of Multiple Sclerosis.

Study 2: Feasibility of home-based FBI for physical and cognitive symptoms of Multiple Sclerosis.

Each study involves a 2-arm, Phase-1, randomized controlled clinical trial to evaluate the effect of FBI on physical, cognitive function, and daily living among people with MS (PwMS). Study 1 is conducted in a lab setting, while Study 2 is conducted at home with additional safety measures. A total of 150 people with multiple sclerosis will be recruited and telephone screened, with an expected enrollment of 120 (60 per phase). After in-person screening, 96 eligible participants (48 per phase) will undergo pre-training assessment and randomization into FBI or Stretching groups. Training sessions will occur twice a week for four months. Anticipating a 15-17% attrition rate, the target sample size is 80 (40 per phase) for completion of the study. Post-training assessments will be conducted after four months to evaluate FBI's impact on physical and cognitive functions. This evidence-based protocol, previously successful with neurological and older adult populations, intends to provide a low-cost, safe, and effective intervention for PwMS in clinical and community settings, including rural areas.

DETAILED DESCRIPTION:
1.0 BACKGROUND/SCIENTIFIC RATIONALE (Study 1 and 2) Of the 1 million adults living with multiple sclerosis (MS) in the United States, over 80% have physical impairment, an estimated 45-60% have cognitive impairment and 20-30% will develop severe dementia. Physical deficits include muscular weakness, spasticity, sensorimotor dysfunction, and imbalance, which co-occur with cognitive dysfunction and directly impact community mobility and overall quality of life. Cognitive deficits include slowed processing speed and reaction time, poor executive functions like planning and problem-solving, and learning and memory deficits. Physical and cognitive deficits rarely remit after onset and are associated with secondary problems with mobility and balance, resulting in increased fall-risk. Whereas treatments targeting restoration of physical function in PwMS have been established, research informing effective management of cognitive dysfunction is in its early stages. Further, there is limited evidence for pharmacological and rehabilitation approaches that can target both physical and cognitive dysfunction. Yet, there have been recent calls for greater focus on unique modes of exercise training as the most promising approach.

Exercise training interventions have yielded modest, but consistent improvements in physical function, walking ability, and fatigue in PwMS. Whereas there is extensive evidence on exercise training targeting physical function, there is comparatively much less known about exercise training targeting cognitive function in PwMS, and this literature is not yet conclusive. Additionally, previous interventions among PwMS have rarely incorporated components of functional balance for treating physical and cognitive dysfunction. Interventions like aerobic and/or strength training are effective in improving physical function, yet effects on cognitive dysfunction might not be very robust. Indeed, cognitive improvements after protocols of aerobic and/or strength-based exercise training might be limited because these modalities might share limited brain resources with physical domains and cognitive tasks, resulting in only a minor transfer of improvements to physical and cognitive performance. On the other hand, there is more evidence of common neural resources shared between cognitive tasks and balance control (e.g., vestibular, visuospatial processing, executive function, attention). Thus, focusing on functional balance training could have a greater activation of the central nervous system (CNS) integrative frameworks for treating cognitive dysfunction in PwMS. It could further have secondary benefits of improving fall efficacy, physical activity, and community mobility thereby mediating change in measures of quality of life among PwMS. Thus, the investigators propose a novel, multicomponent exercise intervention named Functional Balance Intervention (FBI) for improving physical and cognitive function and other measures of daily living among PwMS. The effects of FBI will be tested in a laboratory setting (Study 1) and then tested in a home-based setting (Study 2) in parallel. For both studies, the FBI will be compared to a control group, who will complete an equivalent dosage of stretching. Results from the proposed Phase-I Randomized Controlled Trial (RCT) will inform the research community to launch a line of larger Phase-II RCT examining the comparative effectiveness of the FBI program among PwMS. The findings from this project can also serve as preliminary groundwork for conducting large-scale clinical trials to assess comparative effectiveness of FBI with other pre-established interventions particularly for individuals with restricted mobility and/or restricted access to onsite healthcare services.

2.0 OBJECTIVES (Study 1 and 2) The two-study project is an alternative, non-pharmacological intervention, which represents an important avenue for treating physical and cognitive symptoms of MS and aims to impact measures of mobility and quality of life. Through this project, the investigators will simultaneously examine the effects of FBI compared to stretching among PwMS in a lab-based setting (Study 1) and home-based setting (Study 2). Study 1 and 2 will run in parallel i.e., all data collection, analysis, and dissemination activities will occur simultaneously. For both studies, the investigators first postulate that a Functional Balance Intervention (FBI) can result in immediate improvements in physical function, possibly mediated via improvements in secondary endpoints of dual-task balance, functional mobility, and gait. Secondly, the investigators postulate the possibility that cognition shares more similar neural processes with balance control than with other functional domains, such that CNS adaptations induced by functional balance training could translate into immediate in cognition40. The improvements in physical and cognitive function will mediate improvements in other measures of daily living.

Below are the combined specific aims for Study 1 and 2:

Aim 1: Examine the effect of the FBI (Intervention Group) on physical function in PwMS compared to a stretching program (Control Group).

Hypothesis 1: After 4 months of training, the FBI will show significantly higher improvements in physical function compared to the stretching.

Aim 2: Examine the effect of a multicomponent FBI on cognitive function compared to PwMS in the stretching program.

Hypothesis 2: After 4 months of training, the FBI will show significantly higher improvements in cognitive function compared to the stretching.

Aim 3: Examine the effects of the multicomponent FBI compared to the control group among PwMS on measures of daily living (dual task performance, balance confidence community mobility, and quality of life).

Hypothesis 3: After 4 months of training, the FBI will show significantly higher improvements in measures of daily living compared to stretching.

3.0 Research Design Both sub-studies included in this project (i.e., Study 1 and 2) involve a randomized controlled trial design to establish the feasibility and initial effect of a multicomponent, Functional Balance Intervention (FBI) for immediate improvements in physical and cognitive function, and measures of daily living among persons with multiple sclerosis (PwMS). Study 1 will include training sessions in the lab, and Study 2 will include training sessions at home. Data collection procedures for Study 1 and 2 will run in parallel.

A total sample of 120 participants with Multiple Sclerosis (60 in each study) will be enrolled in this project. The investigators expect ~20% in-person screening failures. Hence, the investigators expect that ~96 PwMS will be eligible to be included in the study, undergo pre-training assessment, and then randomized into 2 groups. The Interventional Group (n=24 for Study 1 and n=24 for Study 2) will undergo a multi component Functional Balance Intervention for 4 months, whereas in the Control Group (n=24 for Study 1 and n=24 for Study 2) will receive a stretching intervention for 4 months.

Study overview (Study 1 and 2) All participants will undergo the following procedures.

* Week 1: Recruitment and phone screening
* Week 2: In-person screening (2 hours)
* Week 3: Pre-training assessment (2 hours)
* Week 4: Random Assignment
* Week 5-20: Training sessions (1 hour/day, 2 times per week for 4 months)
* Week 21: Post-training assessment (2 hours)

ELIGIBILITY:
Inclusion criteria:

Telephone screening (for Study 1 and 2):

* Age group: Adults between 55-80 years of age
* Self-reported diagnosis of Multiple Sclerosis
* Be on stable disease modifying therapy (DMT) for ≥6 months.
* Has not received physical therapy or occupational therapy services for ≥6 months.
* Able to stand up from a chair independently with or without use of handrails.
* Score between 25-75% on the 12-item Multiple Sclerosis walking scale, which indicates that they have mobility disability or walking dysfunction.
* Absence of any other acute or chronic neurological (Stroke, Parkinson's disease), cardiopulmonary, musculoskeletal (injuries like fractures or dislocations or pathologies like Rheumatoid arthritis) or systemic diagnosis, all conditions that except Multiple Sclerosis that can directly impact individual's ability to stand and walk.
* Can understand and communicate in English because the protocol will only be delivered in English.
* Be willing to complete all aspects of the study protocol (outcome assessments, 4-month training, accelerometer wear, etc.).
* Individuals who give a positive response (Yes) to the question of whether the participants feel that their memory or thinking skills worsened lately?" will be marked as potential individuals with mild cognitive impairment.
* Must be willing to come to the lab for 2 times a week for four months for training sessions (for Study 1 participants only).
* Must have access to the internet and must be willing to attend weekly zoom calls and undergo monthly tests on zoom (for Study 2 participants only).
* Must be living with a family member (for Study 2 participants only).
* Must have a helper buddy to be present during the home exercise sessions and monthly progression evaluation Zoom calls with the researcher (for Study 2 participants only).

In-person Screening (for Study 1 and 2):

* Must have mobility Disability, a score of 4.0-6.5 on the Expanded Disability Status Scale (EDSS).
* Must have mild cognitive impairment, a score of 18-25 on the Montreal Cognitive Assessment (MoCA) and score >1 but less than 2.5 standard deviations on 2 or more measures within at least 1 domain (e.g., memory, language, attention/processing speed, executive function, visuospatial abilities) on the established criteria named "Jak / Bondi" criteria.
* Must be physically inactive, a score <14 on the questionnaire named "Godin leisure time" questionnaire.

Exclusion Criteria:

Telephone Screening (for Study 1 and 2):

* MS Relapse or exacerbation ≤3 months
* Recent major surgery (< 6 months) or hospitalization (< 3 months) that might interfere with testing/training.
* Complaints of shortness of breath or uncontrolled pain (>3/10 on visual analogue scale (VAS)) at rest to avoid complications/injuries during testing/training.
* Uncontrolled/untreated hypertension or diabetes to avoid cardiovascular complications during testing/training.
* Self-reported history of bone fracture in the last six months to avoid complications/injuries during testing/training.
* Self-reported disability in performing activities of daily living (with or without assistive device).
* Self-reported diagnosis of epilepsy or uncontrolled seizures in the past year.
* Intake of sedative drugs (diazepam, lorazepam, midazolam, propofol, dexmedetomidine, thiopental) that might interfere with testing/training.
* Intake of any Alzheimer's Disease (AD) or dementia modifying medications (donepezil, rivastigmine, galantamine, aducanumab) as well as other anticipated FDA approved drugs that may be approved during the next 5 years. Individuals who are enrolled in any AD disease modifying drugs trials that might interfere with testing/training or affect the ability to understand instructions will also be excluded.
* Intake of anti-depressants or anxiety drugs.
* Moderate or high risk for possible injury or death when undertaking strenuous or maximal exercise as indicated by reporting a 'YES' on any of the seven items on the Physical Activity Readiness Questionnaire. These participants will be excluded from participation, and further advised to seek medical guidance from their physician.
* People with severe cognitive impairment will be excluded, indicated by a score of 18 or higher on the Telephone Interview for Cognitive status (TICS-M). These participants will be advised to seek medical guidance from the physician.
* Currently undergoing any cognitive rehabilitation for higher brain functions or physical rehabilitation.
* Pacemaker users

In-person Screening (for Study 1 and 2):

* Cardiovascular abnormalities: Heart Rate > 85% of age-predicted maximal heart rate, systolic blood pressure (SBP) > 165 millimetre of mercury (mmHg), diastolic blood pressure > 110 mmHg during rest OR systolic blood pressure < 90 mmHg and/or mean arterial blood pressure < 65 mmHg OR oxygen saturation < 95% during rest.
* Osteopenia (a T - Score of ≤-2.5 on heel ultrasound). Participants with a score ≤ -2.5 will be advised to seek medical guidance from their physician.
* Loss of protective peripheral sensations (inability to perceive 5.07/10 g on the Semmes Monofilament testing).
* Global aphasia (A score of <71% on the Mississippi Aphasia Scoring test)
* Peripheral nerve injuries (traumatic nerve lacerations, pathological nerve damage).
* High fall-risk, <40/56 on Berg Balance Scale (for Study 2 participants only)
* Inability to walk 1 block with or without an assistive device (for Study 2 participants only)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-01-09 (Estimated); Study Completion 2027-01-09 (Estimated)

PRIMARY OUTCOMES:
Change in physical function | Week 3 (Pre-training Assessment), Week 21 (Post-training assessment)
  Physical function will be assessed via the Short Physical Performance Battery (SPPB). This batter includes tests for standing balance and muscle strength and is widely used among older adults and people with multiple sclerosis. Higher scores indicate better performance.
Change in cognitive function | Week 3 (Pre-training Assessment), Week 21 (Post-training assessment)
  Cognitive function will be assessed by the Brief International Cognitive Assessment (BICAMS) The BICAMS is widely used in people with MS and consists of 3 sub-tests including the Symbols Digit Modalities test for assessing processing speed, the California Verbal Learning Test-II for assessing verbal learning and memory and the Brief Visuospatial Memory also for assessing learning and memory as a part of the BICAMS. All these tests are paper pencil questionnaires to assess different domains of cognitive function. Higher scores indicate better performance.
Change in dual task balance performance | Week 3 (Pre-training Assessment), Week 21 (Post-training assessment)
  Dual task balance performance will be assessed via the limits of Stability with the letter number sequencing test. The Limits of Stability test assesses balance on a computerized balance system, which requires participants to shift weight without losing balance. Maximum excursion will be the outcome assessed using the Limits of Stability test. The Letter Number Sequencing test will be performed simultaneously. This test includes cognitive task involving generating alternating number-letter sequences. The accuracy and total responses will be the outcome measures recorded via this test. Higher values for accuracy and responses indicate better performance.
Change in dual task gait performance | Week 3 (Pre-training Assessment), Week 21 (Post-training assessment)
  Dual task gait performance will be assessed via the Timed-up and Go test with the letter number sequencing test. The Timed-up and Go test evaluates functional mobility among individuals with multiple sclerosis. Participants will be asked to stand from a chair, walk 3 meters, and sit back. Lesser time to complete indicates better performance. The Letter Number Sequencing test will be performed simultaneously. This test includes cognitive task involves generating alternating number-letter sequences. The accuracy and total responses will be the outcome measures recorded via this test. Higher values for accuracy and responses indicate better performance
Change in measured community mobility | Week 3 (Pre-training Assessment), Week 21 (Post-training assessment)
  The investigators will use the ActiGraph sensor to assess change in measured community mobility. Participants will be asked to wear the accelerometer device for the following 7 days for at least 12 hours per day. Participants will be asked to always wear the watch except during bathing, charging it, and sleeping. All of these are reliable and sensitive measures for assessing community mobility among people with multiple sclerosis. Greater number of steps per day indicate greater community mobility.
Change in self-reported community mobility | Week 3 (Pre-training Assessment), Week 21 (Post-training assessment)
  The University of Alabama at Birmingham (UAB) has established a paper pencil questionnaire named "Lifespace Scale Questionnaire" will be used to assess change in self-reported community mobility. The Lifespace scale questionnaire measures a person's mobility in five areas: outside the bedroom, outside the house, in the neighborhood, outside of the neighborhood but in town, and outside town during the past four weeks. Higher scores indicate greater community mobility.
Change in self-reported quality of Life | Week 3 (Pre-training Assessment), Week 21 (Post-training assessment)
  This will be assessed using the MS Impact Scale (MSIS-29), a self-reported measure that includes both physical (20 items) and psychological (9 items) aspects of life quality. Higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Change in walking performance | Week 3 (Pre-training Assessment), Week 21 (Post-training assessment)
  Walking performance will be assessed via the the Dynamic Gait Index (DGI). This test examines dynamic balance through various functional tasks performed in daily living and is a commonly used test among individuals with multiple sclerosis. Higher scores indicate better performance.
Change in walking speed | Week 3 (Pre-training Assessment), Week 21 (Post-training assessment)
  Walking endurance will be assessed using the Timed 25-Foot Walk test. This test measures mobility and leg function performance and is a reliable assessment of used commonly among people with multiple sclerosis over time. Lesser time to complete the test indicates better performance.
Change in balance confidence | Week 3 (Pre-training Assessment), Week 21 (Post-training assessment)
  Balance confidence will be assessed using the Activities-Specific Balance Confidence Scale (ABC), which asks individuals to rate their level of confidence (0-100%) that they will not lose their balance while performing various activities of daily living, such as getting onto an escalator or reaching into a cabinet. This measure has also been shown to be reliable for assessing people with multiple sclerosis. Higher percentage scores indicate better confidence.
Change in functional independence | Week 3 (Pre-training Assessment), Week 21 (Post-training assessment)
  Functional independence will be assessed via the Functional assessment measure (FAM). This test is a 12-item assessment measure to assess functional independence among people with Multiple Sclerosis. The items include self-care items, sphincter control, mobility items, locomotion, communication and psychological adjustment and cognitive function. Higher scores indicate more independence.

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi Bhatt, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kannan L, Vora J, Bhatt T, Hughes SL. Cognitive-motor exergaming for reducing fall risk in people with chronic stroke: A randomized controlled trial. NeuroRehabilitation. 2019;44(4):493-510. doi: 10.3233/NRE-182683. PMID 31256084
- [Background] Motl RW, Sandroff BM, Kwakkel G, Dalgas U, Feinstein A, Heesen C, Feys P, Thompson AJ. Exercise in patients with multiple sclerosis. Lancet Neurol. 2017 Oct;16(10):848-856. doi: 10.1016/S1474-4422(17)30281-8. Epub 2017 Sep 12. PMID 28920890
- [Background] Motl RW, Sandroff BM. Benefits of Exercise Training in Multiple Sclerosis. Curr Neurol Neurosci Rep. 2015 Sep;15(9):62. doi: 10.1007/s11910-015-0585-6. PMID 26223831
- [Background] Sandroff BM, Klaren RE, Pilutti LA, Dlugonski D, Benedict RH, Motl RW. Randomized controlled trial of physical activity, cognition, and walking in multiple sclerosis. J Neurol. 2014 Feb;261(2):363-72. doi: 10.1007/s00415-013-7204-8. Epub 2013 Dec 10. PMID 24323244
- [Background] Amato MP, Zipoli V, Portaccio E. Multiple sclerosis-related cognitive changes: a review of cross-sectional and longitudinal studies. J Neurol Sci. 2006 Jun 15;245(1-2):41-6. doi: 10.1016/j.jns.2005.08.019. Epub 2006 Apr 27. PMID 16643953